CLINICAL TRIAL: NCT02886416
Title: Study of Co-adaptation Between Human Immunodeficiency Virus (HIV) and Cluster of Differentiation 8 (CD8) Cellular Immunity, for 27 Years of Natural Evolution and on Treatment
Brief Title: Co-adaptation Between Human Immunodeficiency Virus (HIV) and Cluster of Differentiation 8 (CD8) Cellular Immunity
Acronym: "ImmunoCo27"
Status: Completed | Type: Observational
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: ANRS EP60; 2016-A00400-51 (Other: ANSM)
Record Dates: First submitted 2016-08-29; First posted 2016-09-01 (Estimated); Last update posted 2018-09-28 (Actual); Status verified 2016-09

CONDITIONS: HIV Infection
Keywords: HIV infection
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — frozen PBMC
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Non interventional study

SUMMARY:
The objective is to characterize the viral evolution and viral factors determining HIV virulence, the evolution of the HIV reservoir in PBMC and the co-evolution of anti-HIV CD8 T cell repertoires. The coordinated study of virus evolution, host responses and identification of genetic determinants of virulence should allow to better understand mechanisms of HIV pathogenicity and persistence of mutations in viral reservoirs.

DETAILED DESCRIPTION:
The importance of the still unmet challenges raised by researches on the eradication of the HIV reservoirs and by the need for developing efficient vaccines against HIV, imposes a much deeper understanding the molecular mechanisms regulating the co-evolution and the co-adaptation between HIV and its host during the natural course of the disease an during treatment. The unique cell collection established 27 years ago in an ANRS cohort (ImmunoCo) and the new methods of ultra deep sequencing, or " next generation sequencing", allow to produce innovative analysis of the HIV variability and of reservoirs as well as of the repertoires used by CD8 T cells responses to provide new insights in the very long term relationships between the virus and its host. The objective is to progress at unprecedented levels in the understanding of these mechanisms thanks to the unique opportunity offered by this Immunoco cohort initially composed of 152 patients infected by HIV, most of them untreated when recruited from 1991 to 97 at Pitié-Salpêtrière hospital, with 28 subjects still followed in this hospital and efficiently treated for the last 15 years. The ImmunoCo cohort had initially been set up to study the characteristics of the cytotoxic T lymphocyte (CTL) responses to HIV with disease progression. This exceptional and still available 1991-97 cell collection enriched of extra samples from 1988 to nowadays, allow us to perform a retrospective longitudinal analysis over 27 years in the 28 patients still followed-up, with a new blood sampling in 2016. The project involves 5 highly experienced teams and aims at characterizing in parallel: 1) the viral evolution and viral factors determining virulence, as markers predicting progression of infection, by performing an ultra deep sequencing of the whole HIV genome and of viral variants archived in blood mononuclear cells (PBMC), and 2) the evolution of the reservoir in PBMC and of the distribution of variants archived in those reservoirs over time, in relationship with exposure to the various selective pressures due to CTL or antiretroviral therapy (ART), 3) the co-evolution of anti-HIV CD8 T cell repertoires: the hypothesis is that the emergence of new CD8 T clonotypes displaying a great sensibility for variant antigens, or a cross-reactivity able to recognize similarly wild-type and mutant epitopes allow an efficient long term control of viral replication, and that cell loss by clonal exhaustion is associated to disease progression. The coordinated study of virus evolution, host responses and identification of genetic determinants of virulence should allow to better understand mechanisms of HIV pathogenicity and persistence of mutations in viral reservoirs, especially of defective mutants or resistant mutants to ART, as well as the co-adaptation of CD8 T cell repertoires and of viral variability determining the capacities of viral control by anti-HIV CD8 T cells. Altogether these results should open new strategies for inhibiting viral replication and for controlling viral reservoirs for therapeutic and vaccinal perspectives.

ELIGIBILITY:
Inclusion Criteria:

* Initially included in the ANRS Immunoco cohort and still followed in the Infectious Diseases department by Pr C. Katlama team

Exclusion Criteria:

* None

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients infected with HIV included in the ANRS Immunoco cohort.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Longitudinal study of the co-adaptation of HIV and immune host factors in 28 patients with HIV followed for 27 years. | 27 years

CONTACTS AND LOCATIONS:
Overall Officials: Victor Appay, phD, Principal Investigator — INSERM S1136

IPD SHARING:
Plan to Share IPD: Yes
Scientific publication